CLINICAL TRIAL: NCT07312994
Title: Vegan, Vegeratian, or Omnivore: Dietary Effects on the Brain Tissue Biomarkers
Brief Title: Analysis of NfL and GFAP in Different Dietary Patterns
Status: Recruiting | Type: Observational
Sponsor: Salzburger Landeskliniken (Other)
Collaborators: Medizinische Einrichtungen der Universität Düsseldorf (Unknown); Medizinische Fakultät der Universität zu Köln (Unknown); Universitätsklinkum Münster - Medizinische Klinik und Poliklinik B (Other)
Responsible Party: Principal Investigator, Tobias Moser, apl. Prof., Salzburger Landeskliniken
Other Study IDs: 1119/2025
Record Dates: First submitted 2025-12-09; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Neurofilament Light Chain; Glial Fibrillary Acidic Protein; GFAP; Vegan Diet; Vegetarian Diet
MeSH Terms: conditions — Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Omnivore
- Vegan
- Vegetarian

SUMMARY:
This observational study aims to investigate the impact of different dietary patterns on brain tissue biomarkers in healthy young adults by measuring blood levels of NfL and GFAP.

The primary research question is: Do vegan, vegetarian, or omnivorous diets influence NfL and GFAP levels?

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals who have followed a vegan, vegetarian, or omnivorous diet for at least one consecutive year
* Aged between 18 and 40 years
* Provision of written informed consent

Exclusion Criteria:

* Diagnose neurological disorders (e.g. neurodegenerative, inflammatory, autoimmune, infectious, vascular)
* Eating disorders
* Excessive alcohol consumption
* Pregnancy
* Recent moderate to severe infection (within the past 12 weeks) , including SARS-CoV-2
* Recent trauma, injury, or surgery (within the past 12 weeks)
* Significant BMI fluctuations (>5 points) within the last year
* Patients who have been using Proton pump inhibitors (PPIs) for an extended period (e.g., 1 month).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young and healthy individuals aged between 18 and 40 years
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Blood levels of the following biomarkers: neurofilament light chain (NfL) in pg/mL, glial fibrillary acidic protein (GFAP) in pg/mL. | Once at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Christian-Doppler-Klinik, Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No